CLINICAL TRIAL: NCT03130257
Title: Blood Pressure Checks for Diagnosing Hypertension (BP-CHECK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CER-1511-32979
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Blood Pressure
Keywords: blood pressure measurement
MeSH Terms: interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinic Blood Pressure Measurement (Active Comparator): Participants will be asked to check their blood pressure at their clinic once within the subsequent three weeks.
  Interventions: Diagnostic Test: Clinic Blood Pressure Measurement; Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring (Reference Standard)
- Home Blood Pressure Measurement (Active Comparator): Participants will receive a validated upper-arm home blood pressure monitor and asked to take two measurements in the morning and two in the evening for at least 5 days over three weeks.
  Interventions: Diagnostic Test: Home Blood Pressure Measurement; Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring (Reference Standard)
- Kiosk Blood Pressure Measurement (Active Comparator): Participants will be asked to use a validated blood pressure kiosk in their clinic or local pharmacy to measure their blood pressure three times on three separate days over three weeks.
  Interventions: Diagnostic Test: Kiosk Blood Pressure Measurement; Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring (Reference Standard)

INTERVENTIONS:
Diagnostic Test: Clinic Blood Pressure Measurement — Participants will be asked to check their blood pressure once within the subsequent three weeks.
  Arms: Clinic Blood Pressure Measurement
Diagnostic Test: Home Blood Pressure Measurement — Participants will receive a validated upper-arm home blood pressure monitor and asked to two measurements in the morning and two in the evening for at least 5 days over three weeks.
  Arms: Home Blood Pressure Measurement
Diagnostic Test: Kiosk Blood Pressure Measurement — Participants will be asked to use a validated blood pressure kiosk in their clinic or local pharmacy to measure their blood pressure three times on three separate days over three weeks.
  Arms: Kiosk Blood Pressure Measurement
Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring (Reference Standard) — Participants will be asked to wear an arm cuff and ambulatory blood pressure monitor for 24 hours, with measurements taken every 30 minutes during the day and every 60 minutes at night.

SUMMARY:
Hypertension is usually diagnosed at a clinic or doctor's office when a patient has blood pressure (BP) that is high for several measurements. However, about 30 percent of patients with high BP in clinics have normal BP outside of clinics. This is called white-coat hypertension. Correct diagnosis of hyper-tension is important to prevent strokes, heart attacks, and heart failure but also to avoid making people worry or take medicines when they don't need to.

To avoid misdiagnosis of hypertension, the US Preventive Services Task Force (USPSTF), which makes national recommendations about disease screening, recommends people should have 24-hour BP ambulatory monitoring (i.e., an arm cuff and BP monitor worn for 24 hours, with measurements taken every 30 minutes during the day and every 60 minutes at night), with home BP monitoring over several days as an alternative. However, most patients have never heard of 24-hour BP monitoring, and physicians rarely order it. Physicians sometimes use home BP monitoring, but not according to recommended guidelines. BP kiosks, for example at drug stores, offer another option. Newer models are accurate and easy to use.

BP-CHECK will identify participants, ages 18 to 85, with high BP at their last clinic visit and invite them to a screening visit. Participants with high BP at the screening visit (510 patients) will be randomized and assigned to 1) clinic BP, 2) home BP, or 3) kiosk BP diagnostic groups for confirming a new diagnosis of hypertension. The clinic BP group will have BP measured at one clinic visit. The home BP group will measure BP two times, twice a day, for five days. The kiosk BP group will measure BP three times on three separate days at a kiosk at their clinic or nearby drugstore. Participants will complete their diagnostic tests over approximately three weeks. They will then be asked to complete 24-hour BP monitoring. Participants will complete surveys at baseline prior to randomization, after diagnostic tests, and at six months.

Hypothesis 1: Compared to the reference standard (24-hour BP), home BP and kiosk BP will be more accurate than clinic BP. Hypothesis 2: Participants with clinic, home, or kiosk BP results concordant with reference standard results will prefer home or kiosk to clinic and 24-hour BP. Hypothesis 2: Participants with clinic, home, or kiosk BP results concordant with reference standard results will prefer home or kiosk to clinic and 24-hour BP.

DETAILED DESCRIPTION:
The investigators will compare the accuracy and acceptability (i.e., comfort, convenience) of clinic, home, and kiosk BP testing to 24-hour BP ambulatory monitoring. The investigators will look at the impact of the study on outcomes that matter to participants: their BP and whether participants feel better or worse overall, worry about BP, and change health behaviors (e.g., lowering salt intake).

Our study team includes patients. The study team also has patient and stakeholder advisors to ensure our study is conducted properly and is not a burden to patients and providers. The investigators will share study results with patient participants and publish papers in scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in the health plan for two years, no diagnosis of hypertension in the prior 2 years or more,
* not on anti-hypertensive medications,
* a high blood pressure at their last clinic visit (systolic blood pressure > or equal to 140 mm Hg or diastolic blood pressure > or equal to 90,
* planning to remain a Kaiser Permanente patient for the next six months,
* able to converse and read in English,
* required to have elevated blood pressure at the screening visit (BP taken 2 times, high each time).

Exclusion Criteria:

* children and pregnant women,
* patients with end-stage renal disease,
* dementia,
* atrial fibrillation and other significant arrhythmias.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A final de-identified data set will be made available to the Patient-Centered Outcome Research Institute (PCORI). This data set will include de-identified, individual-level data and meet specifications set by our Institutional Review Board for sharing such data. The analytic data set will include data dictionaries and descriptions of the data such as cohort identification, study participant characteristics, and data captured electronically and via patient surveys. Parties may request data from Dr. Beverly Green and will need to indicate their plans for data use, acknowledge the source of the data in publications, and, if possible, collaborate with BP-CHECK research group.

REFERENCES:
- [Derived] Hansell LD, Hsu CW, Munson SA, Margolis KL, Thompson MJ, Ehrlich KJ, Hall YN, Anderson ML, Evers SC, Marcus-Smith MS, McClure JB, Green BB. Patient Experiences With Blood Pressure Measurement Methods for Hypertension Diagnosis: Qualitative Findings From the BP-CHECK Study. Am J Hypertens. 2024 Oct 14;37(11):868-875. doi: 10.1093/ajh/hpae088. PMID 38995194
- [Derived] Hall YN, Anderson ML, McClure JB, Ehrlich K, Hansell LD, Hsu CW, Margolis KL, Munson SA, Thompson MJ, Green BB. Relationship of Blood Pressure, Health Behaviors, and New Diagnosis and Control of Hypertension in the BP-CHECK Study. Circ Cardiovasc Qual Outcomes. 2024 Feb;17(2):e010119. doi: 10.1161/CIRCOUTCOMES.123.010119. Epub 2024 Feb 8. PMID 38328915
- [Derived] Green BB, Anderson ML, McClure JB, Ehrlich K, Hall YN, Hansell L, Hsu C, Margolis KL, Munson SA, Thompson MJ. Is Hypertension Diagnostic Testing and Diagnosis Associated With Psychological Distress? Am J Hypertens. 2024 Jan 1;37(1):69-76. doi: 10.1093/ajh/hpad083. PMID 37688515
- [Derived] Hsu C, Hansell L, Ehrlich K, Munson S, Anderson M, Margolis KL, McClure JB, Hall YN, Thompson M, Joseph D, Green BB. Primary care physician beliefs and practices regarding blood pressure measurement: results from BP-CHECK qualitative interviews. BMC Prim Care. 2023 Jan 25;24(1):30. doi: 10.1186/s12875-022-01950-1. PMID 36698062
- [Derived] Thompson MJ, Anderson ML, Cook AJ, Ehrlich K, Hall YN, Hsu C, Margolis KL, McClure JB, Munson SA, Green BB. Acceptability and Adherence to Home, Kiosk, and Clinic Blood Pressure Measurement Compared to 24-H Ambulatory Monitoring. J Gen Intern Med. 2023 Jun;38(8):1854-1861. doi: 10.1007/s11606-023-08036-3. Epub 2023 Jan 17. PMID 36650328
- [Derived] Green BB, Anderson ML, Cook AJ, Ehrlich K, Hall YN, Hsu C, Joseph D, Klasnja P, Margolis KL, McClure JB, Munson SA, Thompson MJ. Clinic, Home, and Kiosk Blood Pressure Measurements for Diagnosing Hypertension: a Randomized Diagnostic Study. J Gen Intern Med. 2022 Sep;37(12):2948-2956. doi: 10.1007/s11606-022-07400-z. Epub 2022 Mar 3. PMID 35239109
- [Derived] Green BB, Anderson ML, Campbell J, Cook AJ, Ehrlich K, Evers S, Hall YN, Hsu C, Joseph D, Klasnja P, Margolis KL, McClure JB, Munson SA, Thompson MJ. Blood pressure checks and diagnosing hypertension (BP-CHECK): Design and methods of a randomized controlled diagnostic study comparing clinic, home, kiosk, and 24-hour ambulatory BP monitoring. Contemp Clin Trials. 2019 Apr;79:1-13. doi: 10.1016/j.cct.2019.01.003. Epub 2019 Jan 8. PMID 30634036

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinic Blood Pressure Measurement: Participants will be asked to check their blood pressure at their clinic once within the subsequent 3 weeks.
  Blood Pressure Measurement: We are comparing 3 types of measuring blood pressure for making a new diagnosis of hypertension, clinic blood pressure, home blood pressure, and kiosk blood pressure measurements over a 3 week diagnostic time period
- Home Blood Pressure Measurement: Participants will receive a validated upper-arm home blood pressure monitor and asked to take two measurements in the morning and two in the evening for at least 5 days over 3 weeks.
  Blood Pressure Measurement: We are comparing 3 types of measuring blood pressure for making a new diagnosis of hypertension, clinic blood pressure, home blood pressure, and kiosk blood pressure measurements over a 3 week diagnostic time period
- Kiosk Blood Pressure Measurement: Participants will be asked to use a validated blood pressure kiosk in their clinic or local pharmacy.
  Blood Pressure Measurement: We are comparing 3 types of measuring blood pressure for making a new diagnosis of hypertension, clinic blood pressure, home blood pressure, and kiosk blood pressure measurements over a 3 week diagnostic time period
Period: Overall Study
Arm/Group | Clinic Blood Pressure Measurement | Home Blood Pressure Measurement | Kiosk Blood Pressure Measurement
Started | 172 | 170 | 168
Completed | 171 | 170 | 166
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinic Blood Pressure Measurement | Home Blood Pressure Measurement | Kiosk Blood Pressure Measurement | Total
Number analyzed (Participants) | 172 | 170 | 168 | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 99 | 102 | 304
  >=65 years | 69 | 71 | 66 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.2) | 59.3 (13.2) | 58.9 (12.9) | 58.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 86 | 79 | 247
  Male | 90 | 84 | 89 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 8 | 19
  Not Hispanic or Latino | 160 | 165 | 157 | 482
  Unknown or Not Reported | 4 | 2 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 9 | 10 | 9 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 13 | 13 | 8 | 34
  White | 136 | 137 | 136 | 409
  More than one race | 6 | 4 | 6 | 16
  Unknown or Not Reported | 7 | 4 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 172 | 170 | 168 | 510
Baseline systolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 149.4 (9.8) | 149.9 (11.0) | 150.1 (9.4) | 149.8 (10.1)
Baseline diastolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 88.5 (9.3) | 87.9 (9.2) | 88.0 (9.6) | 88.1 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Comparative Performance of Clinic, Home, and Kiosk
Description: To compare the performance of clinic, home, and kiosk blood pressure to 24-hour blood pressure (reference standard) for new hypertension diagnoses. Our primary outcome is differences in mean systolic and diastolic blood pressure comparing clinic, home, and kiosk to 24-hour BP.
Time Frame: Randomization to three weeks
Population: The primary analysis population included all participants who completed 14 or more daytime 24-hour BP measurements, plus one or more measurements according to their randomization group.
Measure: Mean (95% Confidence Interval); unit: millimeters of mercury
Arm/Group | Clinic Blood Pressure Measurement | Home Blood Pressure Measurement | Kiosk Blood Pressure Measurement
Number analyzed (Participants) | 142 | 152 | 140
millimeters of mercury
  Systolic BP Mean difference diagnostic vs 24-hour | -4.7 [-7.3 to -2.2] | -0.1 [-1.6 to 1.5] | 9.5 [7.5 to 11.6]
  Diastolic BP Mean difference diagnostic vs 24-hour | -7.2 [-8.8 to -5.5] | -0.4 [-1.4 to 0.7] | 5.0 [3.8 to 6.2]
Statistical Analysis 1: Comparison: Clinic Blood Pressure Measurement vs Home Blood Pressure Measurement vs Kiosk Blood Pressure Measurement; We used linear regression models to estimate the mean difference in BP between diagnostic measurement and daytime average 24-hr BP for each randomization group. Models were estimated using generalized estimating equations with robust standard errors, and adjusted for age, sex, BMI, education, and baseline systolic and diastolic BP. Separate models estimated mean differences (diagnostic protocol - 24-hr BP) between groups for systolic and diastolic BP; Test type: Equivalence — The study planned for a sample size of 510 and 80% protocol completion, resulting in sample size 136 per group. With this sample size, the least detectable difference (LDD) is 4.1 mmHg systolic BP (SBP) and 2.8 mmHg diastolic BP (DBP) between any two groups (assuming Standard Deviation 12.1 and 8.3 for SBP and DBP respectively). Actual sample sizes completing protocol were 142, 149, and 111 for Clinic, Home, and Kiosk groups respectively, resulting in LDD of at least 4.3 for SBP and 3.0 for DBP; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: Self-reported adverse events were collected post-randomization via survey at: 1) 3 weeks; 2) 3 weeks and one day (after collection of 24-hour BP monitor data); and 3) 6-months.
Description: The definitions of adverse event or serious adverse event do not differ from ClinicalTrials.gov definitions. Adverse events were collected using an open text self-report question "Since you enrolled in this study, about [x-time] ago, have you experienced any new and serious health problems?" All responses were collated and coded.
Arm/Group | Clinic Blood Pressure Measurement | Home Blood Pressure Measurement | Kiosk Blood Pressure Measurement
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/170 | 0/168
Serious Adverse Events (participants affected / at risk) | 5/172 | 2/170 | 3/168
Other Adverse Events (participants affected / at risk) | 38/172 | 38/170 | 35/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic Blood Pressure Measurement (N=172) | Home Blood Pressure Measurement (N=170) | Kiosk Blood Pressure Measurement (N=168)
Hospitalization: Back operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hospitalization: Surgery for enlarged prostate & bladder stones (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hospitalization: Surgery for removal appendix, bowel resection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hospitalization: Bladder surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hospitalization: Knee replacement surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Severe allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization: Surgery to implant stents (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic Blood Pressure Measurement (N=172) | Home Blood Pressure Measurement (N=170) | Kiosk Blood Pressure Measurement (N=168)
Discomfort, pain, irritation or bruisng from 24-hour monitor (Skin and subcutaneous tissue disorders) | 15 (15) | 5 (5) | 7 (7)
Sleep disruption (General disorders) | 1 (1) | 2 (2) | 2 (2)
Restlessness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 6 (6)
Anxiety (General disorders) | 0 (0) | 3 (3) | 0 (0) — Anxiety generated by using 24-hour BP monitor
High cholesterol (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Flu (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gluten intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (General disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abnormal EKG (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Toe surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
MRSA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Low B12 and iron (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gall stones (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Loss in erection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Swelling of hands, lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Leg/hip injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach flu/nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory track infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pain NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Deteriorating vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid nodules (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Stress (General disorders) | 0 (0) | 0 (0) | 1 (1)
Epigastric parasite infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nerve damage from frostbite (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants had to have high blood pressure (BP) to be eligible, thus our results may not be generalizable to a population with lower BPs. Diverse groups were somewhat under-represented, but reflective of the underlying demographics of the region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03130257/Prot_SAP_000.pdf